CLINICAL TRIAL: NCT01631461
Title: The Prevalence of Yeast and Bacteria in Women With Painful Breastfeeding and the Diagnostic Value of Signs and Symptoms
Brief Title: Painful Breastfeeding and Bacterial or Yeast Infection
Status: Completed | Type: Observational
Sponsor: Göteborg University (Other)
Collaborators: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: PainBreastfeed
Record Dates: First submitted 2012-06-12; First posted 2012-06-29 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Breast Infection
Keywords: pain; breast feeding; yeast; candida albicance; staphylococcus aureus; Signs and symptoms
MeSH Terms: conditions — Mastitis; Pain; Breast Feeding; Staphylococcal Infections; Signs and Symptoms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1. Deep pain group: 1. Deep pain group; Pain in the breast
- 2. Superficial pain group: Pain on the nipple and/or aereola
- 3. Control group: No pain or other breastfeeding problems

SUMMARY:
The aim of this study is to investigate the prevalence of yeast and bacteria in women with breastfeeding pain and to identify signs and symptoms.

DETAILED DESCRIPTION:
Painful breastfeeding is one of the most common reasons for early weaning. Persistent pain associated with breastfeeding can sometimes be difficult to diagnose and is a source of frustration for the breastfeeding women as well as for healthcare providers.

The diagnosis of candida infection in breastfeeding women is generally based on signs and symptoms identified in case reports and without any culture. Breastfeeding pain has been described as superficial or deep in some studies. This deep pain syndrome as caused by candida or bacteria has been questioned. A few studies have cultured breast milk from women with deep breast pain and found Candida albicans infections or bacterial infections usually caused by Staphylococcus aureus. There still remains controversy and lack of evidence for candidiasis affecting the lactating breast as well as bacteria causing the pain. Ensured diagnostic methods are important due to the resistant problem with both antibiotics and antifungals. Only one study has described five key symptoms associated with candida. It was shiny, flaky nipple/areola, burning pain on the nipple/areola, non-stabbing pain or stabbing pain in the breast.

The objective of this study was to investigate the prevalence of candida and bacteria in women with superficial or deep breastfeeding pain and to identify signs and symptoms linked to candida or bacteria in breast milk and nipple/areola.

ELIGIBILITY:
Inclusion Criteria:

* scored pain > = VAS 4

Exclusion Criteria:

* breastfeeding technique problems
* clinical signs of mastitis
* muscular pain
* breast surgery
* use of antibiotic or antifungal treatment during the last preceding week
* temperature > = 37 degree Celsius

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group 1 and 2: Selected from the breastfeeding receptions (n=2) at Sahlgrenska University hospital and Skövde hospital Group 3, controls: Selected from Primary health care clinics
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2006-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Bacteria | Baseline (at admission)
  Occurrence of bacteria: yes/no
Yeast | Baseline (at admission)
  Occurence of yeast: yes/no

SECONDARY OUTCOMES:
Pain | Baseline (at admission)
  VAS
Signs | Baseline (at admission)
  Nipple areola: cracks, red/pink, flaky, shiny, blurred, swollen, itching, smarting
Bacteria at follow-up | 2 weeks after baseline
  Occurence of bacteria: yes/no
Yeast at follow-up | 2 weeks after baseline
  Occurence of yeast: yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Marie Berg, PhD,MPH,MNS, Study Director — Sahlgrenska Academy at University of Gothenburg